CLINICAL TRIAL: NCT03881228
Title: Patient Centered Intervention to Prevent Tuberculosis Among Children Under Five Years Old Who Are Household Contacts of Persons With Tuberculosis
Brief Title: Patient Centered Intervention to Prevent Tuberculosis Among Children Under Five Years Old
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 103161
Record Dates: First submitted 2019-03-14; First posted 2019-03-19 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2022-05

CONDITIONS: Tuberculosis; Pediatric ALL; Behavior, Health
MeSH Terms: conditions — Tuberculosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 1. at enrollment, caretakers will receive an educational booklet for caretakers explaining why IPT needs to be given
  2. at enrollment and weekly for 24 weeks, caretakers will receive a children's storybook, with weekly installments, over the 6-month course of IPT as a non-monetary incentive
  3. weekly, caretakers will receive short messages services (SMS) reminders delivered to the caretaker for the weekly pick-up.
  Interventions: Behavioral: Increasing the completion of IPT
- Standard of care (No Intervention): Routine care at the health facility

INTERVENTIONS:
Behavioral: Increasing the completion of IPT — Behavioral intervention with three components to increase the completion of IPT among children
  Arms: Intervention

SUMMARY:
Isoniazid preventive therapy (IPT) reduces the risk of tuberculosis in 60%. Young children are at higher risk of developing severe forms of TB, though this can be prevented with a full course of IPT. Preliminary data indicate that 60% of eligible children start IPT, and 30% complete it. Furthermore, children can be exposed to more than one case of TB in the household. Adults exposed to TB in the household setting are not necessarily aware of their risk. Uncertainties in the decisions of staff to prescribe IPT and limited health literacy among caretakers and families contribute to this. The investigators will determine the efficacy of an intervention package to increase IPT adherence and completion among children < 5 years old exposed to TB in the household. The investigators will assess the efficacy of the intervention by 1) measuring IPT completion at 6 months after treatment initiation and by 2) determining adherence to IPT by measuring isoniazid in urine at weeks 2, 8 and 24 in a random cluster sample of 10 health facilities and 20 control facilities with 10 children included in each facility (100 in intervention and 200 in control). The investigators will measure fidelity and reach, and acceptability among caretakers and health staff. The intervention package will consist of: 1) educational booklet for caretakers explaining why IPT needs to be given 2) a children's storybook, with weekly installments, over the 6-month course of IPT as a non-monetary incentive and 3) short messages services (SMS) reminders delivered to the caretaker for the weekly pick-up

In September 2020, the protocol was updated to adapt to the COVID19 situation in Lima. One of the secondary outcome (isoniazid concentration in urine) was cancelled and the full intervention (educational booklet, weekly children storybook and weekly SMS) is now delivered through WhatsApp.

DETAILED DESCRIPTION:
A cluster randomized study was designed, randomizing 10 health facilities to the intervention arm and 20 to control arm. In each, 10 children will be recruited. The mother, or the main caretaker in the intervention arm will receive the intervention package: 1) an educational booklet indicating the importance of IPT, adherence to IPT as well as information on how to give it daily for six months. Thereafter, the mother or main caretaker receives 2) a chapter of a children storybook delivered weekly and 3) SMS to remind her of the pick up, as well as weekly SMS containing a motivating message. Until March 2020, component 1 and 2 of the intervention package were delivered in person, since September 2020 and in adaptation to the SARS Cov2 pandemic, these are delivered via WhatsApp. Children in the control arm will receive the standard of care which consists of a advice and counseling given by the doctor and nurse at the health facility.

The investigators will assess the efficacy of the intervention by 1) measuring IPT completion at 6 months after treatment initiation. The secondary outcome originally planned (determining adherence to IPT by measuring isoniazid in urine at weeks 2, 8 and 24) has been cancelled in adaptation to the SARS Cov2 pandemic.

Fidelity, reach and acceptability will be measured among caretakers and staff with an in depth interview at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Caretakers of a child who is 1) < 5 years old 2) contact of a TB patient 3) has an IPT prescription from the TB physician and 4) has a smartphone that can use WhatsApp to receive the intervention.

Exclusion Criteria:

* Caretaker does not want to participate or cannot provide consent

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Isoniazid preventive treatment completion at week 24 recorded in treatment card | 24 weeks
  Completion of 24 weeks of IPT as per weekly pick ups registered in TB forms

SECONDARY OUTCOMES:
Isoniazid preventive treatment completion at week 20 recorded in treatment card | 20 weeks
  Completion of 20 weeks of IPT as per weekly pick ups registered in TB forms
Questionnaire on self reported adherence to daily treatment | 24 weeks
  Self report of providing daily dose IPT to the child at home as reported by the caretaker to the question: did you give the daily dose to the child? possible answers are yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Otero, MD PhD, Principal Investigator — Universidad Peruana Cayetano Heredia
Locations (1):
- Instituto de Medicina Tropical Alexander von Humboldt, Lima, Peru

IPD SHARING:
Plan to Share IPD: Yes
All study data can be shared with other researcher for research purposes as allowed in the IRB application.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Upon completion of the study, for five years.
Access Criteria: Individual patient data will be submitted by the PI (Larissa Otero) upon request by other researchers.

REFERENCES:
- [Derived] Otero L, Zetola N, Campos M, Zunt J, Bayer A, Curisinche M, Ochoa T, Reyes M, Vega V, Van der Stuyft P, Sterling TR. Isoniazid preventive therapy completion in children under 5 years old who are contacts of tuberculosis cases in Lima, Peru: study protocol for an open-label, cluster-randomized superiority trial. Trials. 2023 Jan 24;24(1):54. doi: 10.1186/s13063-022-07062-6. PMID 36694242